CLINICAL TRIAL: NCT05885347
Title: Innovative Teaching Solutions to Improve the Outcomes of Home Caregivers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, José Joaquín Mira Solves, Principal investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI00868
Record Dates: First submitted 2023-03-31; First posted 2023-06-01 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Medication Errors and Other Product Use Errors and Issues
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Placebo Comparator): This caregivers group will not receive any intervention different to the routinely practice.
  Interventions: Other: Control group
- Video Intervention (Experimental): Caregivers will be taught by a video intervention about how to develop their home tasks during an hour.
  Interventions: Other: 360 videos
- Virtual reality (Experimental): Caregivers will be taught by a VR intervention during 20minutes about how to develop their home tasks.
  Interventions: Other: VR
- Augmented reality (Experimental): Caregivers will be taught by a AR intervention during 20minutes about how to develop their home tasks.
  Interventions: Other: AR

INTERVENTIONS:
Other: 360 videos — Caregivers will receive 2h session of 360 videos about caring and medication errors. Then Caregivers will be recorded performed the task worked in 360 videos instantly after the education and after 6 months.
  Arms: Video Intervention
Other: VR — Caregivers will receive 2h session of VR about caring and medication errors. Then Caregivers will be recorded performed the task worked inVR instantly after the education and after 6 months.
  Arms: Virtual reality
Other: AR — Caregivers will receive 2h session of AR videos about caring and medication errors. Then Caregivers will be recorded performed the task worked in AR videos instantly after the education and after 6 months.
  Arms: Augmented reality
Other: Control group — Caregivers will follow the routine and then will be recorded performing their labour as a caregiver after 6 months.
  Arms: Control group

SUMMARY:
Background. Population ageing is leading to an increase in the number of multi-pathological and polymedicated patients. These patients are at increased risk of suffering adverse events due to medication errors (ME), especially if Barthel≤55. The management of their medication places an added burden of stress on those who assume responsibility for their care. This task, due to the existing gender gap, falls more often on women.

Objective. To promote the safe use of medication in the home by those who assume the role of caregivers of these patients.

DETAILED DESCRIPTION:
General objective. The main objective is to investigate whether the provision of care at home by caregivers of of people with multi-pathology and polypharmacy by formal/informal caregivers trained in VR/AR is more efficient formal/informal caregivers trained through VR/AR is more efficient than traditional training.

Secondary objectives are to provide competencies (knowledge, skills and attitudes) that contribute to reducing attitudes) that contribute to reducing caregiver care and medication errors by helping caregivers caregivers, helping beneficiaries to stay at home for as long as possible; and to determine the extent to which and to determine the extent to which AI allows us to continuously update VR training material.

VR training material. This project is in line with the WHO SDG 3. "Ensure healthy lives and promote well-being for all at all ages". It also responds to the WHO Medicines Without Harm challenge. At the national level, this study study reinforces those policies that aim to strengthen the new care economy and reduce the gender equality reduce the gender equality gap (Component 22, 16 June 2021). Specific objectives

1. To create innovative materials to increase the effectiveness of training for formal and informal caregivers through informal and formal caregivers through VR/AR (fully immersive 3D videos).
2. To determine the effectiveness and cost-effectiveness of VR/AR training in caregiving by caregivers.

2. To determine the effectiveness and cost-effectiveness of VR/AR training in the provision of care by formal and informal caregivers and compare it with the outcomes of training using traditional procedures.

outcomes of training using traditional procedures. 3. To analyse the ability of VR/AR to reduce errors in the provision of home-based care and medication by formal and informal caregivers and to compare it with the results of training using traditional procedures.

3. To analyse the ability of RL/RH to reduce errors in the provision of care and medication in the home by formal and informal caregivers.

4. To determine the usefulness of VR/RA in increasing caregivers' self-confidence, considering gender-related factors. 5. Determine the feasibility of combining the analysis of data captured during home care using AI (Deep home care using AI (Deep Learning) and the latest technological developments in VR/AR for smartphones in VR/AR for smartphones - virtual mapping (Arcore 1.24) and AR interaction (LifeAR) - to generate fully immersive generate fully immersive environments for caregiver training. METHODOLOGY Feasibility study of VR/AR/AR/IA applications in the context of caregiver training in three phases

1. qualitative (to collect key information for the development of immersive environments for the key information to develop immersive environments for VR/AR-based interventions), (2) qualitative (to collect key VR/AR-based interventions), (2) experimental (to test the effectiveness of the intervention targeting caregivers (informal and formal), (3) qualitative (to test the effectiveness of the caregivers (informal and formal) to provide safe home-based care, including cost-effectiveness analysis, (3) experimental (to test effectiveness of cost-effectiveness analysis, (3) prototype development to capture and analyse performance of home-based care to
2. development of prototypes to capture and analyse home-based care performance to promote improvements in training programmes through VR/AR.

training programmes through VR/AR.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers currently

Exclusion Criteria:

* Be familiar with disruptive technologies or suffer from vertigo

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in errors by caregivers at home | 6 months
  Caregivers will be recorded in the hospital performing their task in a simulation. All errors performed doing that situation will be counted by professionals who will reproduce that videos.

SECONDARY OUTCOMES:
Chronic Patient Experience Evaluation Instrument-IEXPAC | 6 month
  Questionnaire regarding the experience of the patient care in a chronic situation, with 16 statements, that should be read in the order in which they appear and choose the option that best reflects the opinion. There are no right or wrong answers, it is own personal experience that matters. All statements refer to the last 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Fisabio, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT05885347/Prot_SAP_000.pdf